CLINICAL TRIAL: NCT06404424
Title: Consecutive Hemoperfusion and Therapeutic Plasma Exchange in Adult Patients With Septic Shock
Brief Title: Combined Hemoperfusion and Therapeutic Plasma Exchange for Treatment of Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-2022-08
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; lipopolysaccharide sorption; cytokines apsorbtion; extracorporeal therapy
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Baseline therapy: Patients of group one received standard treatment according to Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021, without the use of blood purification methods.
- Baseline therapy + High-volume plasma exchange (HVPE) + Efferon CT hemoperfusion: Patients of second group received standart treatment, like first group and also high volume plasma exschange procedure and hemoperfusion procedure using Efferon CT device.
  Interventions: Device: Efferon CT
- Baseline therapy + High-volume plasma exchange (HVPE) + Efferon LPS hemoperfusion: Patients of third group received standart treatment, like first group and also high volume plasma exschange procedure and hemoperfusion procedure using Efferon LPS device.
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity.
  This device is routinely used for extracorporeal therapy of sepsis to improve hemodynamic function and abrogate septic shock.
  Plasma exchange procedures will be carried out with a replacement volume of 2 plasma volumes with fresh frozen plasma and albumin solution.
  Each patient is scheduled to undergo two separate hemoperfusions lasting 8-10 hours within 48 hours.
  60 minutes before the start of hemoperfusion, additional administration of antimicrobial drugs is performed, taking into account their elimination during plasma exchange and adsorption
  Groups: Baseline therapy + High-volume plasma exchange (HVPE) + Efferon LPS hemoperfusion
Device: Efferon CT — Efferon CT, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that adsorbs excessive cytokines via its intrinsic porosity.
  This device is routinely used for extracorporeal therapy of "cytokine storm" syndrome in the course of severe SARS-CoV-2.
  Plasma exchange procedures will be carried out with a replacement volume of 2 plasma volumes with fresh frozen plasma and albumin solution.
  Each patient is scheduled to undergo two separate hemoperfusions lasting 8-10 hours within 48 hours.
  60 minutes before the start of hemoperfusion, additional administration of antimicrobial drugs is performed, taking into account their elimination during plasma exchange and adsorption
  Groups: Baseline therapy + High-volume plasma exchange (HVPE) + Efferon CT hemoperfusion

SUMMARY:
Sepsis is a critical burden for a healthcare. From 2000 to 2020, the number of publications and clinical studies on the topic of Sepsis and septic shock on the National Library of Medicine resource The National Center for Biotechnology Information has tripled. Sepsis is a life-threatening condition that causes significant pathophysiological changes in the body. Currently, sepsis is understood as organ dysfunction caused by a dysregulatory response of the macroorganism to infection. A special role in this process belongs to the innate and adaptive immune response.

Despite the trend towards improving survival rates, mortality in sepsis remains high - about 25%, reaching 60% with the development of septic shock.

Extracorporeal therapy, as an adjuvant method of treatment, has been used for more than 30 years, but conducting large randomized studies confirming its effectiveness is associated with a complex of problems, including the extreme heterogeneity of the population of patients with sepsis and septic shock, different etiologies and complex pathogenesis, non-identical pathophysiological pathways of the dominant organ dysfunction in specific time period and degree of its severity.

Goal of the study is to evaluate safety and efficiency of combined hemoperfusion and therapeutic plasma exchange in adult patients with septic shock.

DETAILED DESCRIPTION:
Sepsis is a critical burden for a healthcare. From 2000 to 2020, the number of publications and clinical studies on the topic of Sepsis and septic shock on the National Library of Medicine resource The National Center for Biotechnology Information has tripled. Sepsis is a life-threatening condition that causes significant pathophysiological changes in the body. Currently, sepsis is understood as organ dysfunction caused by a dysregulatory response of the macroorganism to infection. A special role in this process belongs to the innate and adaptive immune response.

Despite the trend towards improving survival rates, mortality in sepsis remains high - about 25%, reaching 60% with the development of septic shock.

Modern understanding of the pathophysiology of sepsis allows us to identify several groups of molecules that are of significant interest as targets for targeted therapy. Activation of Toll-like receptors of neurophils and macrophages by the so-called PAMPs (pathogen-associated molecular patterns) - extracellular bacterial DNA, lipopolysaccharides, flagellin, lipoteichoic acid, peptidoglycan) leads to changes in the transcription of genes involved in the regulation of the inflammatory response, cellular metabolism with a significant release of cytokinessuch as IL-1, TNF-α, IL-2, IL-6, IL-8, IL-10, IFN-γ and complement proteins.

Extracorporeal therapy, as an adjuvant method of treatment, has been used for more than 30 years, but conducting large randomized studies confirming its effectiveness is associated with a complex of problems, including the extreme heterogeneity of the population of patients with sepsis and septic shock, different etiologies and complex pathogenesis, non-identical pathophysiological pathways of the dominant organ dysfunction in specific time period and degree of its severity.

The strategy of using separate methods for extracorporeal elimination of LPS and cytokines yielded controversial results, with an obvious association of endotoxemia and high concentrations of inflammatory mediators with mortality and severity of organ failure.

According to a meta-analysis of Li X et al. 2021, which included 13 RCTs, LPS-selective hemoperfusion was associated with a decrease in mortality, concentration and activity level of endotoxin, and improved hemodynamic parameters. The EUPHAS 2 trial showed the effect of LPS elimination on improvement in hemodynamics, oxygenation and survival, but the nature of the data collection was retrospective, there was no control group, and the study population was highly heterogeneous in the source of infection and severity of the condition. The largest RCT, EUPHRATES, also confirmed an increase in mean arterial pressure and 28-day survival, but only in patients with endotoxin activity levels in the range of 0.6-0.89. The ABDOMIX study did not demonstrate an effect of endotoxin adsorption on mortality and was associated with a large number of technical difficulties during extracorporeal treatment that affected the outcome.

The use of plasma exchange as an integral technique that allows one to simultaneously eliminate both high-molecular toxins and mediators and medium-sized factors seems justified from the point of view of pathogenesis. Many studies have shown a correlation of high VWF levels and low ADAMTS-13 activity in sepsis with mortality, disease severity, and the intensity of both systemic inflammation and disseminated intravascular coagulation. There are similar data for other molecules, the normalization of which by plasma exchange can potentially improve outcome - high levels of NETs, IgA, IgG, d-dimer, PAI-1, C3 and C4 factors of the complement system, and, conversely, low levels of plasminogen, fibrinogen, antithrombin III, protein C are associated with increased mortality. But there is relatively little research on plasma exchange.

Thus, blood purification techniques used for sepsis certainly have a therapeutic effect; it is assumed that their combined use will enhance it, which will potentially improve treatment results.

The need to influence different classes of molecules (weight, kinetics, volume of distribution) of both the immune system and the hemostatic system determines the choice of methods of combined extracorporeal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Sepsis (SEPSIS-3)
* No more than 24 hours from the onset of septic shock.
* Septic shock, defined as hypotension in sepsis:

  1. Persisting after infusion therapy in a volume of 30 ml/kg
  2. Requiring sympathomimetic therapy with one or more of the listed drugs with the indicated doses: norepinephrine - more than 0,05 mcg/kg/min, dopamine - more than 10 mcg/kg/min, adrenaline - more than 0,05 mcg/kg/min,

Exclusion Criteria:

* Inability to achieve and maintain mean arterial pressure more than 65 mm Hg
* History of transfusion reactions, TRALI
* Allergy to heparin, history of HIT
* Uncontrolled bleeding or a high risk of its occurrence
* The presence of cardiovascular events during the last 2 months: AMI, stroke, pulmonary embolism
* Severe congestive CHF
* Terminal CKD, PGD
* HIV infection
* Continuous immunosuppressive therapy
* Severe granulocytopenia (WBC less than 500 cells/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, with clinical signs of septic shock (SEPSIS-3) who were admitted to the intensive care unit (ICU)
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Shock - Free Days | 0-7 days
  All days of life, without vasopressor or inotropic support. A patient is given a value of 0 if they die before day 7 or are still remains in shock at day 7.

SECONDARY OUTCOMES:
ICU - Free Days | 0-60 days
  All days of life spent outside the intensive care unit within 60 days after inclusion in the study. A patient is given a value of 0 if they die before day 60 or are still receiving MV at day 60.
Mechanical ventilation - Free Days | 0-60 days
  All days of life spent without mechanical ventilation. A patient is assigned a value of 0 if he or she dies before day 60 or continues to be on mechanical ventilation on day 60.
Change SOFA score | 0-48 hours
  Value of indicators on the Sequential Organ Failure Assessment (SOFA) Score. Each organ system received a score ranging from 0 (normal) to 4 (most abnormal), with a minimum SOFA score of 0 and a maximum SOFA score of 24.
  The change of SOFA score from baseline (hour 0) at the initiation of hemoperfusion to 48 hours post-treatment initiation.
Change oxygenation index | 0-48 hours
  The change in value of oxygenation index (Pa02 / Fi02) from baseline (hour 0) at the initiation of hemoperfusion to 48 hours post-treatment initiation.
  Oxygenation index (OI) is commonly used to assess the severity of hypoxic respiratory failure (HRF).
  OI < 5 - healthy person; OI 5-25 - indicates lung disease; OI 25-40 - increased mortality; and OI > 40 - consider the use of ExtraCorporeal Membrane Oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Krotenko, PhD, MD, Principal Investigator — City clinical hospital named after S. S. Yudin, Moscow City Health Department
Locations (1):
- City clinical hospital named after S. S. Yudin, Moscow City Health Department, Moscow, Russia